CLINICAL TRIAL: NCT04964219
Title: Analgesic Effects of Low-dose S-ketamine in Patients Undergoing Major Spine Fusion Surgery: A Double-blinded, Randomized Controlled Trial
Brief Title: Analgesic Effects of Low-dose S-ketamine in Major Spine Fusion Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-272
Record Dates: First submitted 2021-07-06; First posted 2021-07-16 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: S-ketamine; Postoperative Analgesia; Spine Fusion
Keywords: S-ketamine; Postoperative Analgesia; Spine Fusion
MeSH Terms: interventions — Esketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S-ketamine group (Experimental): After anesthesia induction, a bolus of 0.15 mg/kg S-ketamine is injected intravenously about 30 min before incision; this is followed by a continuous infusion at a rate of 0.15 mg/kg/h until 1 hour before the end of surgery.
  After surgery, patient-controlled analgesia is provided. The pump is established with S-ketamine 25 mg, dexmedetomidine 100 microgram, and sufentanil 100 microgram, diluted with normal saline to 100 ml. The pump is programmed to deliver 2-ml boluses with a background infusion rate at 1 ml /h and a 10-min lockout interval.
  Interventions: Drug: S-ketamine
- Control group (Placebo Comparator): After anesthesia induction, a bolus of placebo (normal saline) in the same volume is injected intravenously about 30 min before incision; this is followed by a continuous infusion of placebo at the same rate until 1 hour before the end of surgery.
  After surgery, patient-controlled analgesia is provided. The pump is established with placebo, dexmedetomidine 100 microgram and sufentanil 100 microgram, diluted with normal saline to 100 ml. The pump is programmed to deliver 2-ml boluses with a background infusion rate at 1 ml /h and a 10-min lockout interval.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: S-ketamine — After anesthesia induction, a bolus of 0.15 mg/kg S-ketamine is injected intravenously about 30 min before incision; this is followed by a continuous infusion at a rate of 0.15 mg/kg/h until 1 hour before the end of surgery.
  After surgery, patient-controlled analgesia is provided. The pump is established with S-ketamine 25 mg, dexmedetomidine 100 microgram, and sufentanil 100 microgram, diluted with normal saline to 100 ml. The pump is programmed to deliver 2-ml boluses with a background infusion rate at 1 ml /h and a 10-min lockout interval.
  Arms: S-ketamine group
Drug: Placebo — After anesthesia induction, a bolus of placebo (normal saline) in the same volume is injected intravenously about 30 min before incision; this is followed by a continuous infusion of placebo at the same rate until 1 hour before the end of surgery.
  After surgery, patient-controlled analgesia is provided. The pump is established with placebo, dexmedetomidine 100 microgram and sufentanil 100 microgram, diluted with normal saline to 100 ml. The pump is programmed to deliver 2-ml boluses with a background infusion rate at 1 ml /h and a 10-min lockout interval.
  Arms: Control group

SUMMARY:
Despite opioid-based multimodal analgesia, moderate-to-severe pain remains a big problem in patients following multi-segment spinal fusion. As a N-methyl-D-aspartate receptor antagonist, S-ketamine has prominent analgesic effects through activating receptors both in the brain and in the spinal cord, inhibiting the excitatory postsynaptic potential, and thus blunting nociception transmission.

This randomized controlled trial is designed to investigate whether perioperative S-ketamine infusion can decrease pain intensity after major spine fusion surgery.

DETAILED DESCRIPTION:
Multi-segment spinal fusion usually lasts long and produces significant trauma. Patients following this surgery are at high risk of developing moderate-to-severe pain. In a large sample size cohort study investigating pain severity following 179 kinds of surgical procedures, multi-segment spinal fusion ranked the third with a median pain score of 6.6 (assessed with an 11-point scale, where 0=no pain and 10= the worst pain) and a median morphine consumption of 27 mg during the first postoperative day.

High-dose opioids are associated with adverse effects including respiratory depression, sedation, nausea and vomiting, pruritus, and constipation, which are harmful for early postoperative recovery. A previous study showed that about 50% of patients are taking opioids for chronic pain at 3 months after spinal fusion surgery. Chronic pain is considered to be a result of poorly controlled acute postoperative pain. Thus, multimodal analgesia aiming at improving analgesia while decreasing opioid consumption is advocated to control acute postsurgical pain, in order to promote perioperative recovery and prevent chronic pain.

Racemic ketamine, a commonly used N-methyl-D-aspartate receptor antagonist, is a mixture of equal parts of two optical isomers including R-(-)-ketamine and S-(+)-ketamine. It has prominent analgesic effects through activating receptors both in the brain and in the spinal cord, inhibiting the excitatory postsynaptic potential, and thus blunting nociception transmission. Additionally, studies also showed that, when used within the appropriate time, ketamine reduces pain-related sensitization that aggravates postoperative pain. Thus, ketamine is recommended as a part of a multimodal analgesia regimen in clinical practice, especially for patients undergoing major orthopedic surgery. However, the reported psychotropic side effects limit the clinical use of racemic ketamine.

S-ketamine, an S-isomer of ketamine, is twice as potent as the racemic mixture in analgesia, and produces fewer side effects than the racemic ketamine. How, there are only a few studies exploring analgesic effect of S-ketamine in spine fusion surgery. In opioid-dependent patients, Nielsen et al. reported that intraoperative S-ketamine infusion reduced opioid consumption within 24 hours and relieved back pain intensity at 6 months, it also decreased the daily opioid use at 1 year after spinal surgery. On the other hand, the study of Brinck et al. did not found any superiority of intraoperative S-ketamine in reducing oxycodone consumption within 48 hours after lumbar fusion surgery in opioid-naive patients.

Considering these inconsistent results, the effects of S-ketamine in spinal surgery require further clarification. This trial is designed to investigate the analgesic effect of S-ketamine infused both intraoperatively and postoperatively in patients undergoing multi-segment spine infusion surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 80 years.
* Scheduled to undergo multi-segment (≥2) spine fusion surgery.
* Agreed to receive postoperative patient-controlled analgesia.

Exclusion Criteria:

* Refused to participant in this trial.
* Poor blood pressure control in those with hypertension (BP >160/100 mmHg in the ward).
* Previous history of hyperthyroidism or pheochromocytoma.
* Previous history of schizophrenia, epilepsy or Parkinson disease.
* History of sick sinus syndrome, bradycardia (HR <50 beat per min), or atrioventricular block of grade II or higher without pacemaker.
* Severe heart dysfunction (New York Heart Association functional classification 4), hepatic insufficiency (Child-Pugh grade C), renal insufficiency (serum creatinine of 442 μmol/L or above, or requirement of renal replacement therapy), or ASA classification IV or above.
* Unable to complete preoperative assessment due to severe dementia or language barrier.
* Any other conditions that were considered unsuitable for the study participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-05-02 (Actual)

PRIMARY OUTCOMES:
The percentage of patients with moderate-to-severe pain in the first 48 hours after surgery. | Up to 48 hours after surgery
  Moderate-to-severe pain is defined as a numeric rating scale (NRS; an 11-point scale where 0=no pain and 10=the worst pain) pain score ≥4.

SECONDARY OUTCOMES:
Opioid consumption during anesthesia | From induction to end of anesthesia
  Opioid consumption in equivalent-dose of sufentanil
Cumulative opioid consumption after surgery | From end of anesthesia to the 5th day after surgery
  Opioid consumption in equivalent-dose of sufentanil
NRS pain score at rest and with movement | Up to postoperative day 5
  Pain is assessed with a numeric rating scale (NRS; an 11-point scale where 0=no pain and 10=the worst pain)
The percentage of using rescue analgesics | Up to postoperative day 5
  The percentage of using rescue analgesics
Subjective sleep quality | Up to postoperative day 5
  Subjective sleep quality is assessed with NRS scale (0 indicates the best sleep and 10 indicates the worst sleep)
Time to first ambulation | Up to 30 days after surgery
  Time to first ambulation
Quality of recover after surgery | On the third day after surgery
  Quality of recover is assessed with the Quality of Recovery scale, a 15-item Q-15 questionnaire with score ranges from 0 to 150, with higher score indicating better recovery.
Length of hospital stay after surgery | Up to 30 days after surgery
  Length of hospital stay after surgery
The percentage of taking oral analgesics | On the 30th day after surgery
  The percentage of taking oral analgesics
The severity of anxiety and depression | On the 30th day after surgery
  The severity of anxiety and depression is assessed with the Hospital Anxiety and Depression Scale, a 14-item questionnaire with scores range from 0 to 21 for either anxiety or depression. Higher score indicates more severe symptom.
The incidence of postoperative complications and mortality | Up to 30 days after surgery
  The incidence of postoperative complications and mortality

OTHER OUTCOMES:
Sedation or agitation level | Up to 5 days after surgery
  Sedation or agitation was assessed using the Richmond Agitation Sedation Scale (RASS), with scores ranging from -5 (unarousable) to +4 (combative) and 0 indicates alert and calm
The incidence of postoperative nausea and vomiting | Up to 5 days after surgery
  The incidence of postoperative nausea and vomiting
The incidence of delirium | Up to 5 days after surgery
  The incidence of delirium
The incidence of other adverse events (dizziness, nightmares, hallucination and etc.) | Up to 5 days after surgery
  Other adverse events include dizziness, nightmares, hallucination, and others
The percentage of adverse events requiring therapeutic intervention | Up to 5 days after surgery
  The percentage of adverse events requiring therapeutic intervention

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD, PhD, Principal Investigator — Peking University First Hospital
Locations (1):
- Beijing University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233
- [Background] Stein C. New concepts in opioid analgesia. Expert Opin Investig Drugs. 2018 Oct;27(10):765-775. doi: 10.1080/13543784.2018.1516204. Epub 2018 Sep 7. PMID 30148648
- [Background] Connolly J 3rd, Javed Z, Raji MA, Chan W, Kuo YF, Baillargeon J. Predictors of Long-term Opioid Use Following Lumbar Fusion Surgery. Spine (Phila Pa 1976). 2017 Sep 15;42(18):1405-1411. doi: 10.1097/BRS.0000000000002133. PMID 28263225
- [Background] Ocay DD, Li MMJ, Ingelmo P, Ouellet JA, Page MG, Ferland CE. Predicting Acute Postoperative Pain Trajectories and Long-Term Outcomes of Adolescents after Spinal Fusion Surgery. Pain Res Manag. 2020 Feb 24;2020:9874739. doi: 10.1155/2020/9874739. eCollection 2020. PMID 32184913
- [Background] Cozowicz C, Bekeris J, Poeran J, Zubizarreta N, Schwenk E, Girardi F, Memtsoudis SG. Multimodal Pain Management and Postoperative Outcomes in Lumbar Spine Fusion Surgery: A Population-based Cohort Study. Spine (Phila Pa 1976). 2020 May 1;45(9):580-589. doi: 10.1097/BRS.0000000000003320. PMID 31770340
- [Background] Walker CT, Gullotti DM, Prendergast V, Radosevich J, Grimm D, Cole TS, Godzik J, Patel AA, Whiting AC, Little A, Uribe JS, Kakarla UK, Turner JD. Implementation of a Standardized Multimodal Postoperative Analgesia Protocol Improves Pain Control, Reduces Opioid Consumption, and Shortens Length of Hospital Stay After Posterior Lumbar Spinal Fusion. Neurosurgery. 2020 Jul 1;87(1):130-136. doi: 10.1093/neuros/nyz312. PMID 31414128
- [Background] Doan LV, Wang J. An Update on the Basic and Clinical Science of Ketamine Analgesia. Clin J Pain. 2018 Nov;34(11):1077-1088. doi: 10.1097/AJP.0000000000000635. PMID 29927768
- [Background] Brinck EC, Tiippana E, Heesen M, Bell RF, Straube S, Moore RA, Kontinen V. Perioperative intravenous ketamine for acute postoperative pain in adults. Cochrane Database Syst Rev. 2018 Dec 20;12(12):CD012033. doi: 10.1002/14651858.CD012033.pub4. PMID 30570761
- [Background] Park PJ, Makhni MC, Cerpa M, Lehman RA, Lenke LG. The role of perioperative ketamine in postoperative pain control following spinal surgery. J Spine Surg. 2020 Sep;6(3):591-597. doi: 10.21037/jss-19-306. PMID 33102896
- [Background] Avidan MS, Maybrier HR, Abdallah AB, Jacobsohn E, Vlisides PE, Pryor KO, Veselis RA, Grocott HP, Emmert DA, Rogers EM, Downey RJ, Yulico H, Noh GJ, Lee YH, Waszynski CM, Arya VK, Pagel PS, Hudetz JA, Muench MR, Fritz BA, Waberski W, Inouye SK, Mashour GA; PODCAST Research Group. Intraoperative ketamine for prevention of postoperative delirium or pain after major surgery in older adults: an international, multicentre, double-blind, randomised clinical trial. Lancet. 2017 Jul 15;390(10091):267-275. doi: 10.1016/S0140-6736(17)31467-8. Epub 2017 May 30. PMID 28576285
- [Background] Arendt-Nielsen L, Nielsen J, Petersen-Felix S, Schnider TW, Zbinden AM. Effect of racemic mixture and the (S+)-isomer of ketamine on temporal and spatial summation of pain. Br J Anaesth. 1996 Nov;77(5):625-31. doi: 10.1093/bja/77.5.625. PMID 8957979
- [Background] Adams HA, Werner C. [From the racemate to the eutomer: (S)-ketamine. Renaissance of a substance?]. Anaesthesist. 1997 Dec;46(12):1026-42. doi: 10.1007/s001010050503. German. PMID 9451486
- [Background] Pfenninger E, Baier C, Claus S, Hege G. [Psychometric changes as well as analgesic action and cardiovascular adverse effects of ketamine racemate versus s-(+)-ketamine in subanesthetic doses]. Anaesthesist. 1994 Nov;43 Suppl 2:S68-75. German. PMID 7840417
- [Background] Adams HA, Thiel A, Jung A, Fengler G, Hempelmann G. [Studies using S-(+)-ketamine on probands. Endocrine and circulatory reactions, recovery and dream experiences]. Anaesthesist. 1992 Oct;41(10):588-96. German. PMID 1332529
- [Background] Nielsen RV, Fomsgaard JS, Siegel H, Martusevicius R, Nikolajsen L, Dahl JB, Mathiesen O. Intraoperative ketamine reduces immediate postoperative opioid consumption after spinal fusion surgery in chronic pain patients with opioid dependency: a randomized, blinded trial. Pain. 2017 Mar;158(3):463-470. doi: 10.1097/j.pain.0000000000000782. PMID 28067693
- [Background] Nielsen RV, Fomsgaard JS, Nikolajsen L, Dahl JB, Mathiesen O. Intraoperative S-ketamine for the reduction of opioid consumption and pain one year after spine surgery: A randomized clinical trial of opioid-dependent patients. Eur J Pain. 2019 Mar;23(3):455-460. doi: 10.1002/ejp.1317. Epub 2018 Oct 14. PMID 30246357
- [Background] Brinck ECV, Maisniemi K, Kankare J, Tielinen L, Tarkkila P, Kontinen VK. Analgesic Effect of Intraoperative Intravenous S-Ketamine in Opioid-Naive Patients After Major Lumbar Fusion Surgery Is Temporary and Not Dose-Dependent: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial. Anesth Analg. 2021 Jan;132(1):69-79. doi: 10.1213/ANE.0000000000004729. PMID 32167978